CLINICAL TRIAL: NCT00501618
Title: An Open-Label Study Changing Generic Clozapine Formulation to FazaClo® (Clozapine, USP) Orally Disintegrating Tablets in Stable Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Equivalence of Generic Clozapine to Orally Dissolving Clozapine in Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Manhattan Psychiatric Center (Other)
Collaborators: Azur Pharma, Inc (Industry)
Responsible Party: Principal Investigator, Jean-Pierre Lindenmayer, Clinical Director, Manhattan Psychiatric Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 06I/C02-1
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Orally dissolving clozapine; orally disintegrating clozapine; bio-equivalence; desmethylclozapine; clozapine plasma level; equivalence; fazaclo; generic clozapine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fazaclo (Other): open label switch from generic clozapine to Fazaclo
  Interventions: Drug: Fazaclo

INTERVENTIONS:
Drug: Fazaclo — single-arm
  Other Names: Fazaclo clozapine

SUMMARY:
The purpose of this study is to obtain data on equivalence of generic clozapine to Fazaclo (orally disintegrating tablet). Generic clozapine is the most frequently used clozapine and such data is important for clinicians to have.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the equivalence of generic clozapine tablets to FazaClo in patients with schizophrenia or schizoaffective disorder who are already taking generic clozapine and are switched to FazaClo.

In this study, patients receiving a stable twice-daily dose of generic clozapine formulation for the past one month will be switched to FazaClo. A trough steady-state clozapine and desmethylclozapine concentrations will be taken thrice while patient is on generic Clozapine. After the third clozapine level patients will be switched from their generic clozapine formulation to FazaClo, at the same dosage and treatment regimen as the generic clozapine formulation they had been receiving. Trough steady-state clozapine and desmethylclozapine concentration levels will be taken twice, 7 days and 14 days after starting Fazaclo.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) are between 18 and 59 years of age.
* Female patients are not pregnant or breastfeeding and those who are not surgically sterilized, postmenopausal (at least six months), or sexually abstinent are using adequate contraceptive methods (defined as diaphragm, condom, foam/jellies, sponge, and/or oral contraceptives).
* Patients have a diagnosis of 1) treatment-resistant schizophrenia or; 2) schizophrenia, chronic (all types) and in a residual phase or in remission, or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria and are judged to be at chronic risk for reexperiencing suicidal behavior based on history and recent clinical state. In addition, all patients must have a total score on the PANSS of 90 or less.
* Patients have been on a generic clozapine formulation for one month prior to Visit 1 with no changes in clozapine or psychotropic medication dosage in the past one month. Clozapine dose is administered twice daily.
* Patients have no clinically significant abnormalities in the medical history, physical examination, and clinical laboratory tests.
* Patients have given written consent after being advised of the nature and risks of the study and are competent to sign an Informed Consent Form.
* Patients who have shown inconsistent clozapine plasma levels or inconsistent clinical response with a therapeutically adequate daily dose of clozapine as documented in the medical chart or documented by nursing notes about patients' cheeking the oral tablets of clozapine for at least 6 months.

Exclusion Criteria:

* Patients are included in the National Non-Rechallenge Master File for Clozaril.
* Patients have a medical or surgical condition that might interfere with the absorption, metabolism, or excretion of clozapine or FazaClo.
* Patients have a history of granulocytopenia or myeloproliferative disorder, either drug-induced or idiopathic.
* Patients have a total white blood cell (WBC) count below 4000/mm3 or an absolute neutrophil count (ANC) below 2000/mm3.
* Patients have a history of clinically significant cardiovascular, renal, hepatic, respiratory, endocrine (except noninsulin-dependent diabetes mellitus), or gastrointestinal disease.
* Patients have a known history of human immunodeficiency virus infection.
* Patients have a history of epilepsy or seizures or are comatose or experiencing severe central nervous system depression.
* Patients are unable to communicate with the investigator.
* Patients have a history of allergic reactions to clozapine or chemically related psychotropic drugs.
* Patients have a concurrent primary psychiatric or neurological diagnosis, including organic mental disorder (DSM-IV criteria), mental retardation, severe tardive dyskinesia, or idiopathic Parkinson's disease.
* Patients have had electroconvulsive therapy within the past three months.
* Patients have demonstrated clinically significant homicidal behavior within the past 12 months.
* Patients have received an investigational drug within the past 30 days.
* Patients have a history of narrow-angle glaucoma.
* Patients require treatment with drugs that are known to interact with clozapine (e.g., agents having a well-known potential to suppress bone-marrow functioning, drugs that are highly protein-bound, cimetidine, or phenytoin). Clozapine may also potentiate the effects of antihypertensives and anticholinergics; therefore, caution should be taken if patients receiving these drugs are enrolled in the study.
* Patients are morbidly obese (defined as having a body mass index [BMI] greater than 40; BMI = weight [kg]/height [m2]).
* Patients have a known history of phenylketonuria. FazaClo contains aspartame, a source of phenylalanine which can be harmful to patients with phenylketonuria.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the equivalence of generic clozapine tablets to FazaClo in patients with schizophrenia or schizoaffective disorder who are already taking generic clozapine and are switched to FazaClo. | 14 days

SECONDARY OUTCOMES:
Whether side effects are comparable when equivalent plasma levels are present | 14 days
Whether clinical efficacy is maintained after the switch to Fazaclo | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Lindenmayer, MD, Principal Investigator — Manhattan Psychiatric Center; Saurabh Kaushik, MD, Study Chair — Nathan Kline Institute & Manhattan Psychiatric Center
Locations (2):
- United States (2):
  - Manhattan Psychiatric Center, 125th Street, Out Patient Clinic, New York, New York
  - Manhattan Psychiatric Center, Inpatient Unit, New York, New York

REFERENCES:
- See also: Clozapine on Wikipedia — http://en.wikipedia.org/wiki/Clozapine
- See also: Clozapine Registery — http://www.clozapineregistry.com